CLINICAL TRIAL: NCT07286773
Title: Evaluation of the Effectiveness of Biofeedback-Assisted Short Foot Exercises in Individuals With Flexible Pes Planus: A Randomized Controlled Trial
Brief Title: Biofeedback-Assisted Short Foot Exercises in Flexible Flatfoot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Taner Alparslan, Principal Investigator, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0a747ZHs - 2025/689
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pes Planus
Keywords: Flexible Flatfoot; Short Foot Exercise; Biofeedback Training
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BF Group (Experimental)
  Interventions: Other: Biofeedback assisted exercises
- Exerc Group (Active Comparator)
  Interventions: Other: Supervised exercises

INTERVENTIONS:
Other: Biofeedback assisted exercises — Biofeedback-assisted short foot exercise group
  Arms: BF Group
Other: Supervised exercises — Short foot exercise only group
  Arms: Exerc Group

SUMMARY:
The goal of this clinical trial is to compare the effects of biofeedback-assisted short foot exercises and traditional short foot exercises in individuals with flexible pes planus. The study aims to determine whether adding biofeedback to short foot exercises leads to greater improvements in foot biomechanics, balance, and functional ability.

The main questions it aims to answer are:

Does biofeedback-assisted short foot exercise improve plantar pressure distribution and foot posture more than traditional short foot exercise? Does the use of biofeedback result in greater improvements in balance and functional ability? Researchers will compare a biofeedback-assisted short foot exercise program to a traditional short foot exercise program to evaluate their effects on plantar pressure distribution, foot posture, balance, ankle range of motion, and functional outcomes.

Participants will:

Be randomly assigned to either a traditional short foot exercise group or a biofeedback-assisted short foot exercise group Participate in a supervised exercise program twice per week for 6 weeks Complete pre- and post-intervention assessments, including plantar pressure analysis, balance tests, foot posture evaluation, and self-reported functional questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participants aged 18 to 45 years
* Diagnosis of flexible pes planus
* No history of surgery, fracture, or psychiatric disorder

Exclusion Criteria:

* Diagnosis of rigid pes planus
* Age younger than 18 years or older than 45 years
* History of psychiatric disorder or lower extremity trauma

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-10-22 (Estimated)

PRIMARY OUTCOMES:
The Foot and Ankle Ability Measure (FAAM) | Baseline
  The Foot and Ankle Ability Measure (FAAM) is a validated, self-reported questionnaire designed to assess functional limitations associated with foot and ankle conditions. It consists of two subscales: Activities of Daily Living (ADL) and Sports.
  Each item is scored on a 5-point Likert scale, ranging from 0 (unable to perform) to 4 (no difficulty). The total score for each subscale is converted to a percentage, with higher scores indicating better functional ability.
  The FAAM has been shown to be reliable, valid, and responsive to clinical change in individuals with musculoskeletal impairments of the foot and ankle.
The Foot and Ankle Ability Measure (FAAM) | 6 week
  The Foot and Ankle Ability Measure (FAAM) is a validated, self-reported questionnaire used to assess functional limitations associated with foot and ankle conditions. It consists of two subscales: Activities of Daily Living (ADL) and Sports.
  Each item is scored on a 5-point Likert scale, ranging from 0 (unable to perform) to 4 (no difficulty). Total scores for each subscale are converted to percentage scores, with higher values indicating better functional performance.
  The FAAM has demonstrated good reliability, validity, and responsiveness to clinical change in individuals with musculoskeletal impairments of the foot and ankle.
Pedobarographic Analysis | Baseline
  Pedobarographic analysis is an objective method used to assess plantar pressure distribution and contact area during static standing or walking. Measurements are obtained using a computerized pressure platform that records static and dynamic foot loading patterns in real time.
  During the assessment, participants stand or walk barefoot on the pedobarographic platform. The system measures the magnitude and distribution of plantar pressures and contact area across different regions of the foot, including the heel, midfoot, and forefoot.
  This analysis provides quantitative data on load symmetry, pressure distribution, and medial-lateral balance, which are key indicators of foot biomechanics and medial longitudinal arch function.
Pedobarographic Analys | 6 Week
  Pedobarographic analysis is an objective method used to assess plantar pressure distribution and contact area during static standing and walking. Measurements are obtained using a computerized pressure platform that records static and dynamic foot-loading patterns in real time.
  During the assessment, participants stand or walk barefoot on the pedobarographic platform. The system measures the magnitude and distribution of plantar pressures and contact area across different regions of the foot, including the heel, midfoot, and forefoot.
  This analysis provides quantitative data on load symmetry, pressure concentration, and medial-lateral balance, which are important indicators of foot biomechanics and medial longitudinal arch function.

SECONDARY OUTCOMES:
Active Range of Motion | Baseline
  Active ankle range of motion, including plantarflexion and dorsiflexion, will be measured according to the guidelines described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer.
Active Range of Motion | 6 week
  Active ankle range of motion, including plantarflexion and dorsiflexion, will be measured in accordance with the guidelines of the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer.
FPI-6 (Foot Posture Index-6) | 6 Week
  The Foot Posture Index (FPI-6) is a clinical assessment tool used to evaluate static foot posture. It consists of six observational criteria: talar head palpation, curvature above and below the lateral malleolus, calcaneal position in the frontal plane, prominence of the talonavicular joint, height and congruence of the medial longitudinal arch, and forefoot abduction/adduction.
  Each item is scored on a 5-point scale ranging from -2 (indicating supination) to +2 (indicating pronation), resulting in a total score ranging from -12 to +12.
  Lower scores indicate a more supinated foot posture, whereas higher scores indicate a more pronated foot posture. A score close to zero represents a neutral foot alignment.
  Interpretation of Scores
  * 12 to -5: Highly supinated
  * 4 to -1: Slightly supinated
    0 to +5: Neutral
    * 6 to +9: Pronated
    * 10 to +12: Highly pronated
Navicular Drop Test | Baseline
  The Navicular Drop Test is a clinical assessment used to evaluate the degree of medial longitudinal arch collapse by measuring the difference between non-weight-bearing and weight-bearing positions of the foot.
  During the test, the vertical height of the navicular tuberosity from the floor is measured in both a seated (non-weight-bearing) and a standing (weight-bearing) position using a ruler or digital caliper. The difference between these two measurements, expressed in millimeters (mm), represents the navicular drop value.
  A greater navicular drop value indicates increased pronation and lowering of the medial longitudinal arch, whereas smaller values suggest a more neutral or supinated foot posture.
  Outcome Metric
  Difference in navicular height (mm) between seated and standing positions
  Interpretation of Results
  < 5 mm: Minimal or no arch drop (supinated tendency)
  5-9 mm: Normal range
  ≥ 10 mm: Excessive pronation / flatfoot tendency
Y-Balance Test | Baseline
  The Y-Balance Test is a dynamic balance assessment tool used to evaluate an individual's ability to maintain postural control while reaching in multiple directions. The participant stands on one leg at the center of a Y-shaped grid and reaches as far as possible with the contralateral leg in three directions: anterior, posteromedial, and posterolateral. The maximum reach distance for each direction is measured in centimeters (cm) and normalized to leg length to reduce inter-individual variability.
  The test is performed on both lower extremities, and the mean of three successful trials in each direction is recorded. Greater reach distances indicate better dynamic balance performance, whereas shorter reach distances or asymmetry between limbs may indicate balance deficits.
  Outcome Metrics:
  Reach distance (cm) in the anterior, posteromedial, and posterolateral directions Composite Y-Balance Score (%) = [(Anterior + Posteromedial + Posterolateral) / (3 × Limb length)] × 100
FPI-6 (Foot Posture Index-6) | Baseline
  The Foot Posture Index (FPI-6) is a clinical assessment tool used to evaluate static foot posture. It consists of six observational criteria: talar head palpation, curvature above and below the lateral malleolus, calcaneal position in the frontal plane, prominence of the talonavicular joint, height and congruence of the medial longitudinal arch, and forefoot abduction/adduction.
  Each item is scored on a 5-point scale, ranging from -2 (indicating supination) to +2 (indicating pronation), resulting in a total score ranging from -12 to +12.
  Lower scores indicate a more supinated foot posture, whereas higher scores indicate a more pronated foot posture. A score close to zero represents a neutral foot alignment.
  Interpretation of Scores
  * 12 to -5: Highly supinated
  * 4 to -1: Slightly supinated
    0 to +5: Neutral
    * 6 to +9: Pronated
    * 10 to +12: Highly pronated
Y-Balance Test | 6 Week
  The Y-Balance Test is a dynamic balance assessment tool used to evaluate an individual's ability to maintain postural control while reaching in multiple directions. The participant stands on one leg at the center of a Y-shaped grid and reaches as far as possible with the contralateral leg in three directions: anterior, posteromedial, and posterolateral. The maximum reach distance for each direction is measured in centimeters (cm) and normalized to leg length to reduce inter-individual variability.
  The test is performed on both lower extremities, and the mean of three successful trials in each direction is recorded. Greater reach distances indicate better dynamic balance performance, whereas shorter reach distances or asymmetry between limbs may indicate balance deficits.
  Outcome Metrics
  Reach distance (cm) in the anterior, posteromedial, and posterolateral directions Composite Y-Balance Score (%) = [(Anterior + Posteromedial + Posterolateral) / (3 × Limb length)] × 100
Navicular Drop Test | 6 week
  The Navicular Drop Test is a clinical measurement used to assess the degree of medial longitudinal arch collapse by comparing the foot in non-weight-bearing and weight-bearing positions.
  During the test, the vertical height of the navicular tuberosity from the floor is measured in both a seated (non-weight-bearing) and a standing (weight-bearing) position using a ruler or digital caliper. The difference between these two measurements, expressed in millimeters (mm), represents the navicular drop value.
  A greater navicular drop value indicates increased pronation and lowering of the medial longitudinal arch, whereas smaller values suggest a more neutral or supinated foot posture.
  Outcome Metric
  Difference in navicular height (mm) between seated and standing positions
  Interpretation of Results
  < 5 mm: Minimal or no arch drop (supinated tendency)
  5-9 mm: Normal range
  ≥ 10 mm: Excessive pronation / flatfoot tendency

CONTACTS AND LOCATIONS:
Overall Officials: Taner ALPARSLAN, PT, Master's student, Principal Investigator — Istanbul University - Cerrahpasa; Sezen KARABÖRKLÜ ARGUT, Asst. Prof. Dr., Principal Investigator — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul University-Cerrahpaşa, Istanbul, Büyükçekmece
  - Department of Orthopedics and Traumatology, Istanbul Faculty of Medicine, Istanbul University, Istanbul, Fatih

IPD SHARING:
Plan to Share IPD: Undecided